CLINICAL TRIAL: NCT05410457
Title: Study on the Effect of Different Treatment Strategies on Prognosis of Acute Ischemic Stroke(AISDTS)
Brief Title: Different Treatment Strategies on Prognosis of Acute Ischemic Stroke(AISDTS)
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: AISDTS
Record Dates: First submitted 2022-05-26; First posted 2022-06-08 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; clincial indicators; thrombolysis; thrombectomy; neuroimaging; genetics; one-stop multimodal-MRI; stroke related complications
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were collected from routine blood sample.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- thrombolysis group: Inclusion criteria: a) age ≥18 years; B) hospital admission for acute ischemic stroke; C) the time from onset to admission ≤ 4.5 hours; D) received intravenous thrombolysis; E) signed informed consent.
- thrombectomy group: Inclusion criteria: a) age ≥18 years; B) hospital admission for acute ischemic stroke; C) the time from onset to admission ≤ 24 hours; D) vascular assessment by CTA or multimodal MRI; E) received thrombectomy; F) signed informed consent.
- stent group: Inclusion criteria: a) age ≥18 years; B) hospital admission due to ischemic stroke; C) vascular assessment by CTA or multimodal MRI; D) received stent implantation ; E) Signed informed consent.
- regular treatment group: Inclusion criteria: a) age ≥18 years; B) hospital admission due to ischemic stroke; C) received regular medical treatment; D) signed informed consent.
- young stroke group: Inclusion criteria: a) age between 18 and 50 years of age (45/55Y); B) hospital admission due to ischemic stroke; C) received CT or MRI imaging assessment; D) signed informed consent.
- unexplained stroke group: Inclusion criteria: a) age ≥18 years; B) hospital admission due to ischemic stroke; C) Received CT or MRI imaging assessment; D)TOAST was classified as unknown cause type (including two or more causes and no cause was found by auxiliary examination); E) signed informed consent.

SUMMARY:
AISDTS is a prospective registry study, in which clinical information, examination and imaging data of patients with acute ischemic stroke receiving different treatment strategies were collected, grouped and statistically analyzed, and corresponding clinical prediction models were constructed to explore the role of clinical biological indicators in the occurrence and development of stroke.

DETAILED DESCRIPTION:
1. To study which variable or variables (various clinical biological indicators) affect the prognosis of ischemic stroke patients;
2. To study the differences in variables (various clinical evaluations, biological indicators, etc.) among patients receiving different treatment strategies (including thrombolysis group, thrombectomy group, stent group, chronic occlusion reperfusion group and regular treatment group);
3. To study hemoglobin, mean erythrocyte volume, white blood cell count, neutrophil count, lymphocyte count, monocyte count, IL-2, IL-4, IL-6, IL-10, IFNγ, TNFα, C-reactive protein, serum iron and iron-related proteins (ferritin, transferrin, fibromodulin, ceruloplasmin), uric acid, amino acid, lipoprotein, homocysteine, vitamin D and other clinical indicators that correlated with acute ischemic stroke patients and different treatment groups were compared;
4. To study the relationship between blood pressure changes at multiple time points from admission to discharge and clinical manifestations and prognosis of stroke patients, and to make comparison between groups;
5. To study the relationship between ischemic stroke and other variables (clinical assessment, biological, genetic and neuroimaging) in different pathological types;
6. To study the correlation between neuroimaging indicators and clinical evaluation, biomolecular, genetic and other variables;
7. DNA and RNA were extracted from peripheral blood samples of patients with acute stroke for genetic related studies to explore the genetic susceptibility of young stroke and unexplained stroke;
8. To study the role of one-stop multimodal-MRI in the assessment and diagnosis of patients with acute ischemic stroke;
9. To study the adverse reactions (hemorrhage, embolus shedding, gastrointestinal ulcer) and stroke-related complications under different treatment strategies (including thrombolysis group, thrombectomy group, stent group, chronic occlusion reperfusion group and regular treatment group);
10. To study the effect of Sanbexin® (Edaravone and Dexborneol Concentrated Solution for Injection) on inflammation and the prognosis in ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* A) ≥18 years of age; B) hospital admission for ischemic stroke; C) Signed informed consent.

Exclusion Criteria:

* A) patients with incomplete clinical information; B) hospitalization observation time less than 24 hours; C) recent trauma, severe inflammation, severe liver and kidney dysfunction, progressive malignance and other serious diseases; D) baseline mRS score>2; E) informed consent is not signed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital for ischemic stroke were enrolled.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2027-06-24 (Estimated); Study Completion 2027-06-24 (Estimated)

PRIMARY OUTCOMES:
To assess the changes of prognosis of stroke patients under different treatment strategies | 3 months, 6 months, 12 months or 24 months
  assessed by The Modified Rankin Score (mRS) of stroke patients [mild to wores ranging from 0 to 5, 6 represents death].
To assess the early neurological changes of ischemic stroke | 7 days or 14 days
  change from baseline National Institute of Health stroke scalescore (NIHSS) [higher scores mean worse conditions]7 days or 14 days

SECONDARY OUTCOMES:
To assess the incidence of recurrent stroke under different treatment strategies | 7 days-24 months
  record and analyze the incidence of recurrent stroke from 7 days-24 months
To assess the types and incidence of adverse events of ischemic stroke patients | 3 days-24 months
  adverse reactions (hemorrhage, embolus shedding, gastrointestinal ulcer) and stroke-related complications under different treatment strategies
To assess the correlation of RNA/DNA and age factor in acute ischemic stroke | 3 months
  DNA and RNA extracted from peripheral blood samples
To assess the therapeutical effects of Edaravone dexborneol on inflammation and prognosis after acute ischemic stroke | 3 months
  The Modified Rankin Score score (mRS) of stroke patients [mild to wores ranging from 0 to 5, 6 represents death].

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China